CLINICAL TRIAL: NCT05238324
Title: A Phase 1 Open-Label Dose Escalation Study to Evaluate the Safety and Efficacy of HMI-203 in ERT-Treated Adults With Mucopolysaccharidosis Type II (MPS II) (juMPStart Trial)
Brief Title: Safety and Efficacy of HMI-203 in ERT-Treated Adults With MPS II
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Homology Medicines has discontinued development of this program.
Sponsor: Homology Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMI-203-101
Record Dates: First submitted 2021-12-07; First posted 2022-02-14 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Mucopolysaccharidosis II
Keywords: MPS II; Hunter syndrome
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HMI-203 Low Dose Level Cohort 1 (Experimental)
  Interventions: Biological: Genetic HMI-203
- HMI-203 Intermediate Dose Level Cohort 2 (Experimental)
  Interventions: Biological: Genetic HMI-203
- HMI-203 High Dose Level Cohort 3 (Experimental)
  Interventions: Biological: Genetic HMI-203

INTERVENTIONS:
Biological: Genetic HMI-203 — HMI-203 delivered intravenously

SUMMARY:
Phase 1, open-label, sequential ascending dose-escalation study. Designed to evaluate the safety and efficacy of a single IV infusion of investigational gene therapy HMI-203. Males, ages 18 to 45 years inclusive, with MPS II (Hunter syndrome) currently receiving idursulfase ERT (or the equivalent) are eligible to participate. Participants will be followed for safety and efficacy for 5 years.

DETAILED DESCRIPTION:
This Phase 1 study will evaluate the safety and efficacy of HMI-203 gene therapy in adult male participants with MPS II currently being treated with standard-of-care idursulfase ERT or equivalent. Participants will receive a single dose of HMI-203 administered intravenously. There are 3 planned dose cohorts which will consist of 3 participants each.

Entry into the first dose cohort will be separated by a 60-day dosing interval between each participant to allow the Homology Medicines medical monitor to review safety and efficacy data prior to the second and third participants being enrolled. Enrollment of subsequent participants, in cohorts 2 and 3, will be separated by a 21-day dosing interval between each participant for review of safety and efficacy data.

Escalation to the next dose cohort will occur after 21 days of safety, efficacy, and biomarker data have been reviewed by the Homology Medicines independent DMC.

This entire study is comprised of 5 years, with the most frequent follow up visits occurring in the first year.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult males 18-45 years of age at the time of informed consent
* Has capacity and is able to understand the purpose and risks of the study and is willing, able and committed to comply with all study procedures for the duration of the trial (a total of 5 years after gene therapy administration)
* Diagnosis of MPS II based on historically decreased I2S enzyme activity and elevated urine GAGs and/or presence of hemizygous IDS pathogenic variant
* Kaufman Brief Intelligence Test-Second Edition (KBIT2) score ≥ 80
* Compliance with regular treatments of ERT for MPS II for at least 12 months prior to enrollment
* Clinically stable relative to urinary GAG levels, ambulation, and cardiopulmonary status for 12 months preceding enrollment

Key Exclusion Criteria:

* Multiple sulfatase disorder as determined by abnormal activity of another lysosomal sulfatase
* Unresponsive and/or intolerant to idursulfase treatment
* History of BMT, stem cell transplant, or gene therapy
* Presence of anti-capsid neutralizing antibodies
* ALT or AST > ULN; Total or Direct bilirubin > ULN
* International normalized ratio (INR) >1.2 ULN
* Hematology values below the normal range
* Hemoglobin A1c ≥ 6.5% or fasting glucose ≥126 mg/dL
* Contraindication to corticosteroid or tacrolimus use
* Any condition that would not allow the potential participant to complete follow-up examinations during the course of the study or, in the opinion of the investigator, makes the potential participant unsuitable for the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence and severity of treatment emergent adverse events (TEAEs) after a single dose administration of HMI-203 (at each dose level) in adult participants with MPS II | Baseline through 260 weeks
  The following events are defined as TEAEs;
  1. Elevation in serum transaminases (concentration that is > 1.5× ULN) and/or
  2. Elevation in serum direct bilirubin (concentration that is > 1.5× ULN)
Evaluate the incidence and severity of adverse events of special interest (AESIs) after a single dose administration of HMI-203 (at each dose level) in adult participants with MPS II | Baseline through 260 weeks
  The following events are defined as AESIs;
  1. Elevation in serum transaminases (concentration that is > 1.5× ULN) and/or
  2. Elevation in serum direct bilirubin (concentration that is > 1.5× ULN)
Evaluate the effect of HMI-203 single administration on urinary GAG levels within each dose cohort | Baseline to week 52
  Single urine sample GAG levels
Evaluate the effect of HMI-203 single administration on plasma I2S activity within each dose cohort | Baseline to week 52
  Measure trough I2S plasma activity

SECONDARY OUTCOMES:
Evaluate the long-term effect of HMI-203 single administration on plasma I2S activity and concentration within each dose cohort | week 52 to week 260
  Measure trough I2S plasma activity and measure trough I2S plasma concentration
Evaluate the long-term effect of HMI-203 single administration on urinary GAG levels within each dose cohort | week 52 to week 260
  Single urine sample GAG levels
Evaluate the effect of HMI-203 on use of ERT | Baseline through week 260
  Incidence of ERT discontinuation by 52 weeks following HMI-203 administration and among participants who have discontinued ERT by 52 weeks. Annualized frequency of ERT infusions at weeks 24, 52, 76, 104, 156, 208 and 260.
Changes from baseline in 6-minute Walk Test (6MWT) performance | Baseline to timepoints between Week 52 to Week 260
  Change from baseline in mean 6-minute walk test (6MWT)
Changes from baseline in cardiac mass | Baseline; weeks 52, 104, 156, 208, and 260
  Cardiac mass will be evaluated by performing a transthoracic 2-dimensional echocardiogram.
Changes from baseline in cardiac function | Baseline; weeks 52, 104, 156, 208, and 260
  Cardiac function will be evaluated by performing a transthoracic 2-dimensional echocardiogram with doppler flow.
Changes from baseline pulmonary function by evaluating spirometry with lung volumes for FEV1 (Forced Expired Volume). | Baseline; weeks 52, 104, 156, 208, and 260
Changes from baseline pulmonary function by evaluating spirometry with lung volumes for FVC (Forced Vital Capacity). | Baseline; weeks 52, 104, 156, 208, and 260
Changes from baseline pulmonary function by evaluating spirometry with lung volumes for TLC (Total Lung Capacity). | Baseline; weeks 52, 104, 156, 208, and 260
Changes from baseline pulmonary function by evaluating spirometry with lung volumes for RV (Residual Volume). | Baseline; weeks 52, 104, 156, 208, and 260
Changes from baseline pulmonary function by evaluating spirometry with lung volumes for TV (Tidal Volume all in L). | Baseline; weeks 52, 104, 156, 208, and 260
Changes from baseline pulmonary function by evaluating spirometry with lung volumes for FEV1/FVC ratio (Forced Expiry Volume in 1 second/Forced Vital Capacity). | Baseline; weeks 52, 104, 156, 208, and 260
Changes from baseline pulmonary function by evaluating spirometry by DLCO (Diffusing Capacity of the Lungs for Carbon Monoxide mL/min/mmHg). | Baseline; weeks 52, 104, 156, 208, and 260
Change in CSF levels of heparan sulfate | Baseline; weeks 52, 260
  Measure CSF heparan sulfate
Change in CSF levels of dermatan sulfate | Baseline; weeks 52, 260
  Measure CSF dermatan sulfate
Change in CSF levels I2S activity and concentration | Baseline; weeks 52, 260
  Measure CSF I2S activity and concentration
Determine immune response to the HMI-203 delivery capsid by evaluating the incidence of antibodies | Baseline; weeks 52 and 260
  Measurement of anti-AAVHSC antibodies (total and neutralizing)
Determine immune response to iduronate 2-sulfatase enzyme (I2S) | Baseline; weeks -1, 1, 4, 8, 12, 24, 52, 78, 104, and 260
  Measurement of anti-I2S antibodies (total and neutralizing)
Determine immune response via cytotoxic T-lymphocyte CD8+ (ELISpot) | Baseline; week 52

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Utah Pediatric Genetic & Metabolism Clinic, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia
- M.A.G.I.C. Clinic, Ltd., Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No